CLINICAL TRIAL: NCT07206524
Title: Effect of Modifying Magnesium Concentration in Citrate-enriched Dialysate on Hemodialysis-associated Thromboinflammation: a Local Pilot OMAGOD Plus Trial
Brief Title: Effect of Modifying Magnesium Concentration in Citrate-enriched Dialysate on Hemodialysis-associated Thromboinflammation
Acronym: pilot OMAGOD +
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: University of Rochester (Other); Vrije Universiteit Brussel, Jette, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 25113_PILOTOMAGOD
Record Dates: First submitted 2025-09-04; First posted 2025-10-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Hemodialysis; Thromboinflammation; Hemodialysis Complication; End Stage Renal Disease (ESRD)
Keywords: hemodialysis; thromboinflammation; neutrophil extracellular trap formation; dialysate composition; cellular activation; transcriptome analysis
MeSH Terms: conditions — Thromboinflammation; Kidney Failure, Chronic | interventions — Magnesium

STUDY DESIGN:
Intervention Model Description: This study focuses on the additional collection of biological samples during the pilot OMAGOD trial. The original study design-a prospective, randomized, single-blind, parallel-group crossover study-will remain unchanged other than the collection of additional samples. Sample collection for this study will be conducted exclusively at our center and will take place during the last hemodialysis session of each treatment period (3 HD sessions per participant).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acetic acid dialysate (0.5 mmol/L Mg) (Active Comparator): Standardized hemodialysis treatments 3x4hours/week. Intervention: 2 weeks (six hemodialysis sessions) during which patients will be dialyzed with standard acetate-based dialysate containing 0,5 mmol/L magnesium.
  Interventions: Other: Hemodialysis using acetic acid dialysate with magnesium 0.5 mmol/L
- Citric acid dialysate (Mg 1.0 mmol/L) (Active Comparator): Standardized hemodialysis treatments 3x4hours/week. Intervention: 2 weeks (six hemodialysis sessions) using a citric acid dialysate containing magnesium 1.0 mmol/L
  Interventions: Other: Hemodialysis using dialysate containing citric acid and magnesium at a concentration of 1.0 mmol/L
- Citric acid dialysate (Mg 0.75 mmol/L) (Active Comparator): Standardized hemodialysis treatments 3x4hours/week. Intervention: 2 weeks (six hemodialysis sessions) using a citrate-enriched dialysate containing magnesium 0.75 mmol/L
  Interventions: Other: Hemodialysis using citric acid dialysate with magnesium 0.75 mmol/L

INTERVENTIONS:
Other: Hemodialysis using dialysate containing citric acid and magnesium at a concentration of 1.0 mmol/L — Change dialysate compositions being used during hemodialysis treatment in each arm.
  Arms: Citric acid dialysate (Mg 1.0 mmol/L)
Other: Hemodialysis using acetic acid dialysate with magnesium 0.5 mmol/L — Standard dialysate containing acetic acid and magnesium at a concentration of 0.5 mmol/L, used during hemodialysis sessions.
  Arms: Acetic acid dialysate (0.5 mmol/L Mg)
Other: Hemodialysis using citric acid dialysate with magnesium 0.75 mmol/L — Dialysate containing citric acid and magnesium at a concentration of 0.75 mmol/L, used during hemodialysis sessions.
  Arms: Citric acid dialysate (Mg 0.75 mmol/L)

SUMMARY:
This clinical trial investigates whether the composition of dialysate influences hemodialysis-associated thromboinflammation. Specifically, it evaluates the effects of magnesium concentration and acid type in dialysate on immune cell activation and thromboinflammatory responses.

Patients participating to the multicentric pilot OMAGOD trial will be invited to participate to this monocentric plus study.

In the pilot OMAGOD trial, participants will undergo standard hemodialysis (3 sessions/week, 4 hours each) and receive three different dialysate compositions in a crossover design. Each treatment phase lasts two weeks (six sessions).

For the local plus study, during selected sessions (3 per patient - midweek hemodialysis session of the last week of a treatment period), blood samples will be collected (at baseline, hourly, and at the end of dialysis) and additionally, after each session, the used dialysis circuit will be rinsed to recover adherent cells.

The study aims to:

* Assess whether the dialysate composition influences leukocyte and platelet activation .
* Evaluate whether the dialysate composition influences neutrophil extracellular trap (NET) formation.
* Identify novel biomarkers of thromboinflammation using transcriptomic analysis of immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Participants to the OMAGOD pilot trial

Exclusion Criteria:

* Patients who are not participating in the OMAGOD pilot trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Differences in leukocyte counts in rinse fluids of discarded hemodialysis circuit in relation to the dialysate composition | Midweek dialysis session during the final week of each treatment period - week 3 (session 9), week 5 (session 15), week 7 (session 21)
  The primary endpoint will be the difference in leukocyte counts in rinse fluids of discarded hemodialysis circuits in relation to the dialysate composition (acetic acid vs. citric acid Mg 0.75 mmol/L vs. citric acid 1.0 mmol/L)

SECONDARY OUTCOMES:
differences in platelet counts in rinse fluids of discarded hemodialysis circuits in relation to the dialysate composition | Midweek dialysis session during the final week of each treatment period - week 3 (session 9), week 5 (session 15), week 7 (session 21)
  differences in platelet counts in rinse fluids of discarded hemodialysis circuits in relation to the dialysate composition, evaluated by hematologic cell analyzer
Differences in leukocyte and platelet activation markers in blood and rinse fluid samples of discarded hemodialysis circuits measured by flow cytometry in relation to dialysate composition | Midweek dialysis session during the final week of each treatment period - week 3 (session 9), week 5 (session 15), week 7 (session 21)
  differences in leukocyte and platelet activation markers in blood samples and rinse fluids of discarded hemodialysis circuits in relation to the dialysate composition; assessed by mean fluorescence intensity and the relative number of positive cells for the respective activation marker measured by flow cytometry.
Differences in coagulation activation and inflammatory biomarkers measured by multiplex-based immunoassays in relation to dialysate composition | Midweek dialysis session during the final week of each treatment period - week 3 (session 9), week 5 (session 15), week 7 (session 21)
  Biological evaluation of systemic coagulation activation and inflammation in relation to dialysate composition. Biomarkers will be measured using multiplex-based immunoassays from plasma samples collected during midweek dialysis sessions.
Differences in Neutrophil Extracellular Trap (NET) formation in relation to the dialysate composition | Midweek dialysis session during the final week of each treatment period - week 3 (session 9), week 5 (session 15), week 7 (session 21)
  Quantification of NET biomarkers in blood and rinse fluids in relation to the dialysate composition.

CONTACTS AND LOCATIONS:
Overall Officials: Florine Janssens, Medical doctor, Principal Investigator — (1)Department of Nephrology and Arterial Hypertension, Universitair Ziekenhuis Brussel (UZ Brussel), Brussels, Belgium. (2) Kidney diseases, dialysis & transplantation Research Unit (NIER), Vitality Research Group, Vrije Universiteit Brussel (VUB)
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided